CLINICAL TRIAL: NCT05626101
Title: Safety and Efficacy of Scheduled Intravesical Gemcitabine Versus Intravesical BCG for Intermediate and High Risk Non Muscle Invasive Bladder Cancer: A Prospective, Randomized Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gemcitabin vs BCG
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inravesical BCG (Active Comparator): Intravsical induction and maintenance BCG injections.
  Interventions: Drug: BCG
- Inravesical Gemcitabin (Active Comparator): Intravsical induction and maintenance gemcitabin injections.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: BCG — Intravsical induction and maintenance BCG injections.
  Arms: Inravesical BCG
Drug: Gemcitabine — Intravsical induction and maintenance gemcitabin injections.
  Arms: Inravesical Gemcitabin

SUMMARY:
About 40%-80% of NMIBC recur within 6-12 months when managed with TURBT alone, and 10%-25% of the patient's progress to muscle invasive disease. Intravesical therapy enables delivery of high local concentrations of a therapeutic agent within the bladder, which could potentially destroy viable tumor cells that remain following TURBT

DETAILED DESCRIPTION:
Bladder cancer (BC) is the tenth most commonly diagnosed cancer worldwide. Approximately 75% of patients with BC present with disease confined to the mucosa (stage Ta or CIS) or submucosa (stage T1); for younger patients (<40 year) this Percentage is even higher (Babjuk et al., 2022).

About 40%-80% of NMIBC recur within 6-12 months when managed with TURBT alone, and 10%-25% of the patient's progress to muscle invasive disease. Intravesical therapy enables delivery of high local concentrations of a therapeutic agent within the bladder, which could potentially destroy viable tumor cells that remain following TURBT (Ye Z, et al., 2018 and Daneshmand et al., 2022).

The Intravesical BCG injection can reduce the recurrence rate by about 30-40%. For intravesical therapy, chemotherapy drugs such as mitomycin C, gemcitabine, and epirubicin can be used post-TURBT, which is a good alternative treatment for BCG or a second-line treatment (Ansari et al., 2022).

The BCG vaccine was firstly developed by Albert Calmette over a hundred years ago. Its effect on bladder cancer was proposed by Dr. Alvaro Morales about forty years ago. In 1990, BCG was approved by the Food and Drug Administration (FDA) for the treatment of NMIBC and then became the first-line drug in NMIBC up to now (Ansari et al., 2022).

Due to worldwide shortage of BCG, there is a clinical need to develop novel intravesical agents and application forms in order to improve the oncological outcomes in non-muscle invasive bladder cancer (NMIBC). Gemcitabine has been investigated in various clinical trials. It has proven to be superior to BCG re-challenge and mitomycin (MMC) in BCG-unresponsive high-risk NMIBC (Gakis, 2022).

Gemcitabine is a nucleoside analogue with cytotoxic activity mediated by inhibition of DNA synthesis followed by cell apoptosis. The majority of trials examining gemcitabine have been in the setting of prior BCG failure (Balasubramanian et al., 2022).

NMIBC represents a significant global therapeutic challenge, particularly in the era of international BCG shortage due to manufacturing issues. Induction and maintenance intravesical BCG remains the historical gold standard for patients with intermediate or high-risk NMIBC. However, clinicians may be forced to consider alternatives given the current BCG shortage. Attempts to rationalize its use, including dose frequency reduction, have resulted in inferior outcome. Accordingly, there is considerable interest worldwide in assessing alternate approaches to improve oncologic outcomes for patients with NMIBC (Balasubramanian et al., 2022).

The majority of trials examining gemcitabine have been in the setting of prior BCG failure. To our knowledge there are only four trials evaluating initial intravesical gemcitabine without prior BCG usage. Porena et al., 2010 included only 32 patients; Bendary et al. 2011 included 40 patients; Gontero et al., 2013 included 61 patients and Prasanna et al., 2017 included 51 patients. Depending on this fact, we need a well-designed prospective trial including a large number of patients with reasonable follow-up period to estimate the actual benefits and hazards of intravesical gemcitabine injection.

ELIGIBILITY:
Inclusion Criteria:

* The study will include moderate and high risk patients with NMIBC. Very high risk NMIBC patients, whom refusing radical cystectomy.

Exclusion Criteria:

* Active UTI.
* Suspected bladder perforation.
* Hematuria.
* Any contraindications for gemcitabin therapy; hypersenstivity, pregnancy, an infection, hemolytic uremic syndrome, , anemia, decreased blood platelets, low levels of a type of white blood cell called neutrophils.
* Patients whom previously received any inravesical therapy (e.g. prior BCG).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | 2 YEARS
  time from the commencement of induction treatment to recurrence. All recurrences will be confirmed by cystoscopic guided biopsy and histology.
Progression free survival (PFS) | 2 YEARS
  progression in the initial tumour staging during follow-up cystoscopy. All progressions will be confirmed by histopathologic evaluation.

SECONDARY OUTCOMES:
Side effects of intravesical gemcitabine injection. | 2 YEARS
  Side effects of intravesical gemcitabine injection will be measures according to the " Common Terminology Criteria for Adverse Events (CTCAE)" Version 5.0 Published on November 27, 2017 by the U.S. department of health and human services
Side effects of intravesical BCG injection. | 2 YEARS
  Side effects of intravesical BCG injection will be measures according to the " Common Terminology Criteria for Adverse Events (CTCAE)" Version 5.0 Published on November 27, 2017 by the U.S. department of health and human services

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Fawzy Salman, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No